CLINICAL TRIAL: NCT07168083
Title: The Efficacy and Safety of Sacituzumab in Patients With Ovarian Clear Cell Carcinoma After the Progression of Immunotherapy: A Prospective Real-world Study
Brief Title: Efficacy and Safety of Sacituzumab in Patients With OCCC After Immunotherapy Progression
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jing Li, professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2025-526-01
Record Dates: First submitted 2025-08-31; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Cancer; Antibody-drug Conjugates; Clear Cell Adenocarcinoma of Ovary
Keywords: Ovarian Clear Cell Carcinoma; antibody-drug conjugate
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sacituzumab Group: The patient received 5 mg/kg of Sacituzumab per two weeks.

SUMMARY:
Ovarian clear cell carcinoma (OCCC) is a relatively rare but highly malignant epithelial ovarian cancer, accounting for 5%-10% of all ovarian cancers. The incidence of this tumor has significant racial disparity, with the highest incidence in Asians, accounting for 25% of ovarian cancer patients, while in European and American ovarian cancer patients, it only accounts for 4.8%. Due to the unique biological behavior of OCCC, it responds poorly to traditional platinum-based chemotherapy regimens, and the prognosis of patients with advanced and recurrent disease is extremely poor.

OCCC has low sensitivity to platinum-based chemotherapy, especially in recurrent or persistent disease, and the objective response rate (ORR) of chemotherapy is usually less than 10%. Although immunotherapy has shown good results in OCCC, 60% of patients still cannot shrink their tumors after using combination regimens, and 50% of patients will still progress after 6.9 months of treatment. The question of how to treat OCCC after progression on immunotherapy remains a pressing issue. Sacituzumab (SKB264) is an antibody-drug conjugate (ADC) consisting of a humanized anti-trophoblast cell surface antigen 2 (Trop-2) monoclonal antibody conjugated to T030. In the KL264-I-01 study (which included patients with OCCC) in patients with recurrent ovarian cancer, single-agent Sacituzumab achieved an objective response rate of 40%, superior to conventional chemotherapy, with manageable toxicity. OCCC patients who progress on immunotherapy face a dilemma of limited treatment options. Based on this current situation and the potential activity of Sacituzumab the investigators propose Sacituzumab as an option for patients with OCCC after immunotherapy progression.

DETAILED DESCRIPTION:
Ovarian clear cell carcinoma (OCCC) is a relatively rare but highly malignant epithelial ovarian cancer, accounting for 5%-10% of all ovarian cancers. The incidence of this tumor has significant racial disparity, with the highest incidence in Asians, accounting for 25% of ovarian cancer patients, while in European and American ovarian cancer patients, it only accounts for 4.8%. Due to the unique biological behavior of OCCC, it responds poorly to traditional platinum-based chemotherapy regimens, and the prognosis of patients with advanced and recurrent disease is extremely poor.

OCCC has low sensitivity to platinum-based chemotherapy, especially in recurrent or persistent disease, and the objective response rate (ORR) of chemotherapy is usually less than 10%. The OCCC tumor microenvironment indicates that OCCC is a "hot tumor," suggesting that patients may benefit from immunotherapy. This benefit has been confirmed in clinical studies. Although immunotherapy has shown good results in OCCC, 60% of patients still cannot shrink their tumors after using combination regimens, and 50% of patients will still progress after 6.9 months of treatment. The question of how to treat OCCC after progression on immunotherapy remains a pressing issue. Sacituzumab (SKB264) is an antibody-drug conjugate (ADC) consisting of a humanized anti-trophoblast cell surface antigen 2 (Trop-2) monoclonal antibody conjugated to T030. In the KL264-I-01 study (which included patients with OCCC) in patients with recurrent ovarian cancer, single-agent Sacituzumab achieved an objective response rate of 40%, superior to conventional chemotherapy, with manageable toxicity. OCCC patients who progress on immunotherapy face a dilemma of limited treatment options. Based on this current situation and the potential activity of Sacituzumab the investigators propose Sacituzumab as an option for patients with OCCC after immunotherapy progression.

The investigators plan to conduct a prospective, real-world clinical study to enroll patients with OCCC who have developed resistance to immunotherapy and receive Sacituzumab (5 mg/kg intravenous infusion, 2 weeks of treatment). The investigators will prospectively observe and collect treatment responses, efficacy data, and safety events, and compare the efficacy with that of a historical cohort of immunotherapy-resistant patients who received traditional chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed ovarian clear cell carcinoma
* Patients who have progressed on imaging assessment after receiving immunotherapy, including anti-PD-1, PD-L1, and PD-1/PD-L1+CTLA4, and subsequently received Sacituzumab.
* At least one measurable lesion as assessed by RECIST, version 1.1.
* Life expectancy ≥ 12 months.
* Normal renal an liver function, no myelosuppression.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score (PS score) 0-1.
* Participants must have recovered from all toxicities resulting from previous treatment (recovery to < grade 1 or protocol-specified inclusion criteria, based on a CTCAE 5.0 assessment), excluding alopecia.
* Participants must be willing to participate in the study, be compliant, sign the informed consent form, and be able to adhere to protocol-specified visits and procedures.

Exclusion Criteria:

* Receipt of more than two lines of therapy after progression on immunotherapy.
* Previous use of irinotecan or ADCs containing topoisomerase I inhibitors.
* Presence or history of (non-infectious) interstitial lung disease (ILD) or non-infectious pneumonitis requiring steroid treatment
* Documented severe dry eye syndrome, severe meibomian gland disease and/or blepharitis, or a history of corneal disease that prevents delayed corneal healing.
* Concomitant incomplete or complete intestinal obstruction, intestinal fistula of any grade, hydronephrosis that cannot be resolved with a ureteral stent, inflammatory bowel disease or brain metastases.
* Organ transplant recipient.
* ≥ Grade 3 venous embolism
* Active infectious disease of any grade, including tuberculosis.
* Previous history of pelvic or abdominal radiation therapy to any site.
* Concurrent with other types of malignant tumors.
* Mental status abnormalities.
* Pregnant or lactating women; or patients of childbearing potential (male or female) who are unable to use effective medical contraception during the study period and for 6 months after the end of dosing.
* Any other condition deemed inappropriate for participation in this study by the investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study enrolled patients with pathologically diagnosed OCCC who had progressed after treatment with immune checkpoint inhibitors, including anti-PD-1, PD-L1, and PD-1/PD-L1+CTLA4, and subsequently received ruconazole (regardless of the number of lines of therapy received prior to immunotherapy).
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 2 years
  The proportion of patients whose tumor volume was reduced by more than 30% and maintained for 4 weeks

SECONDARY OUTCOMES:
Adverse event | 2 years
  Any adverse events that occur during drug treatment
Overall survival | From enrollment to 2 years after treatment completion
  Time from enrollment to death from any cause
Progression free survival | From enrollment to 2 years after treatment completion
  Time from enrollment to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, Doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Takano M, Sugiyama T, Yaegashi N, Sakuma M, Suzuki M, Saga Y, Kuzuya K, Kigawa J, Shimada M, Tsuda H, Moriya T, Yoshizaki A, Kita T, Kikuchi Y. Low response rate of second-line chemotherapy for recurrent or refractory clear cell carcinoma of the ovary: a retrospective Japan Clear Cell Carcinoma Study. Int J Gynecol Cancer. 2008 Sep-Oct;18(5):937-42. doi: 10.1111/j.1525-1438.2007.01158.x. Epub 2007 Dec 13. PMID 18081792
- [Background] Sugiyama T, Kamura T, Kigawa J, Terakawa N, Kikuchi Y, Kita T, Suzuki M, Sato I, Taguchi K. Clinical characteristics of clear cell carcinoma of the ovary: a distinct histologic type with poor prognosis and resistance to platinum-based chemotherapy. Cancer. 2000 Jun 1;88(11):2584-9. PMID 10861437
- [Background] Gadducci A, Multinu F, Cosio S, Carinelli S, Ghioni M, Aletti GD. Clear cell carcinoma of the ovary: Epidemiology, pathological and biological features, treatment options and clinical outcomes. Gynecol Oncol. 2021 Sep;162(3):741-750. doi: 10.1016/j.ygyno.2021.06.033. Epub 2021 Jul 8. PMID 34247767